CLINICAL TRIAL: NCT01997541
Title: Insertion Depth Comparison of Tracheal Tubes
Status: Completed | Type: Observational
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Jong-Man Kang, Associate professor, Kyung Hee University Hospital at Gangdong
Other Study IDs: Kang528
Record Dates: First submitted 2013-07-15; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Intubation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- plain tube
- reinforced tube

SUMMARY:
There will be a difference of the insertion depth between the types of the endotracheal tube.

ELIGIBILITY:
Inclusion Criteria:

* undergoing surgery under general anesthesia -

Exclusion Criteria:

* upper airway or pulmonary problems
* neck and/or chest distortion
* patients at risk for pulmonary aspiration of gastric content -

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: American Society of Anesthesiologists physical status I, II patients scheduled for elective surgery with general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
the distance between endotracheal tube tip and carina | within 1 minute after intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea